CLINICAL TRIAL: NCT05356845
Title: Oral Health, Orofacial Function and Oral Health Care in Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Merete Bakke, Professor, University of Copenhagen
Other Study IDs: OralHelseParkinson
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Parkinsonian Disorders
MeSH Terms: conditions — Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva and tongue plaque
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD group
- Control group

SUMMARY:
Introduction: Problems with oral health (dental and oral diseases) as well as orofacial function (jaw opening, chewing and salivation problems) are significant challenges for many people with Parkinson's disease (PD). These challenges may be painful, disabling, and cause great psychosocial strain and negatively affect quality of life. Furthermore, they may contribute to an unsecure and unhealthy aging, because eating and enjoyment of food is important for both the physical and psychological wellbeing for elderly and chronically ill patients. It seems that patients with PD often find it difficult to maintain adequate oral hygiene and fail to visit the dentist, which in the end contributes to tooth loss, eating problems, poorer nutrition, social challenges and reduced quality of life.

To be able to plan interventions on a larger scale more detailed knowledge and mapping is necessary on the extent of various manifestations of PD in the orofacial area, the affect on the patients and their quality of life, and how the disease develops in the orofacial area for the patient group over time. The study will clarify the challenges and problems that patients with PD have due to their disease in terms of dental and oral health and function of mouth and jaws. Such information is important both for single patients with respect to prevention and intervention and for development of community health strategies.

Purpose

* to investigate specific orofacial, non-motor and motor symptoms and functions as well as the oral microbiome in patients with PD compared to a control group.
* to examine the quality of life related to oral health in the abovementioned groups.
* to provide information on the orofacial problems in PD for the benefit of single patients with respect to prevention and intervention and for development of community health strategies.

Hypotheses: It is expected that

* patients with PD have more orofacial functional problems and poorer oral health than a control group without PD, and patients with late PD have more orofacial functional problems and poorer oral health than patients with early PD.
* patients with PD have an altered oral microbiome compared to a control group without PD, which possibly may assist in the staging of PD.
* patients with PD have poorer oral health related quality of life and home dental care than a control group without PD.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be able to understand the participant information and must be able to collaborate in connection with the study. Must be able to transport himself to and from the Dental School and must be able to sit upright in a dental chair during the examination.
* Inclusion criteria for patients with PD: Participants must be in stable and well-medicated treatment and affiliated with the Department of Neurology at Bispebjerg Hospital (outpatient clinic N30).
* Inclusion criteria for controls: Persons with comparable age and gender distribution without PD diagnosis.

Exclusion Criteria:

- For all participants: Participants with the diagnosis Sjogren's syndrome, implanted electronic devices in the body (pacemaker, DBS and the like) and / or participants who receive or have received radiation in the head / neck region in connection with cancer treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at the Department of Neurology at Bispebjerg Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Electromyographic analysis | Basline
  Measurment: micro volt. Electromyographic measurement of the resting, chewing, swallowing, jaw opening and teeth clenching of the temporalis muscle, the digastric muscle and the masseter bilaterally. Detected with bipolar surface electrodes during 10 s resting and posture activity, chewing 10 g apple, swallowing 2 mL water, maximal jaw opening and teeth clenching.

SECONDARY OUTCOMES:
Maximum molar bite force | basline
  Measure the maximum molar bite force using a transducer in Newton
Oral related quality of life | baseline
  Oral Health Impact Profile questionnaire with 14 questions regarding disability, pain, discomfort, physical impairment, mental impairment, social impairment and disability. Scale from 0-56
Oral and dental health | Basline
  Measurment: DMFT. Obtained by dental examination and Panoramic radiograph
Nordic Orofacial Test - Screening | Basline
  Meaure of The orofacial function on a scale from 0 to 12

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baram S, Thomsen CE, Ozhayat EB, Karlsborg M, Bakke M. Orofacial function and temporomandibular disorders in Parkinson's Disease: a case-controlled study. BMC Oral Health. 2023 Jun 12;23(1):381. doi: 10.1186/s12903-023-03051-6. PMID 37308874